CLINICAL TRIAL: NCT00790907
Title: FondaparinUx Trial With Unfractionated Heparin (UFH) During Revascularization in Acute Coronary Syndromes (ACS) (FUTURA). A Prospective Study Evaluating the Safety of Two Regimens of Adjunctive Intravenous UFH During PCI in High Risk Patients With Unstable Angina/Non ST Segment Elevation Myocardial Infarction (UA/NSTEMI) Initially Treated With Subcutaneous Fondaparinux and Referred for Early Coronary Angiography (OASIS 8)
Brief Title: Fondaparinux Trial With Unfractionated Heparin (UFH) During Revascularization in Acute Coronary Syndromes (ACS)
Acronym: FUTURA/OASIS 8
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 108888
Record Dates: First submitted 2008-11-13; First posted 2008-11-14 (Estimated); Results first posted 2011-06-07 (Estimated); Last update posted 2017-03-23 (Actual); Status verified 2017-03

CONDITIONS: Acute Coronary Syndrome
Keywords: Unstable angina; Non ST elevation myocardial infarction; PCI; unfractionated heparin; fondaparinux; acute coronary syndrome
MeSH Terms: conditions — Acute Coronary Syndrome; Angina, Unstable; Non-ST Elevated Myocardial Infarction | interventions — Heparin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Open label fondaparinux background and standard dose UFH (Experimental): Subjects indicated for PCI and randomized to receive standard dose UFH
  Interventions: Drug: fondaparinux background and standard dose UFH
- Open label fondaparinux background and low dose UFH (Experimental): Subjects indicated for PCI and randomized to receive low dose UFH
  Interventions: Drug: Fondaparinux background and low dose heparin
- Open label fondapaparinux (Other): Subjects not indicated for PCI and not randomized
  Interventions: Drug: Open label fondaparinux

INTERVENTIONS:
Drug: fondaparinux background and standard dose UFH — Open label fondaparinux syringes pre-filled with 2.5 mg, administered s.c. once daily for up to 8 days or hospital discharge, whichever was earlier. Participants indicated for PCI were randomized to receive adjunctive blinded standard dose UFH (based on planned glycoprotein [GP] IIb/IIIa inhibitor use: 60 units/kilogram (U/kg); no planned use: 85 U/kg and adjusted based on activated clotting time (ACT) [maximum two additional bolus doses]). Participants who presented in the catheterization laboratory and who were receiving commercially available fondaparinux prescribed for the initial treatment of UA/NSTEMI may have been considered for randomization.
  Arms: Open label fondaparinux background and standard dose UFH
Drug: Fondaparinux background and low dose heparin — Open label fondaparinux syringes pre-filled with 2.5 mg, administered s.c. once daily for up to 8 days or hospital discharge, whichever was earlier. Participants indicated for PCI were randomized to receive adjunctive blinded low-dose UFH (50 U/kg), which was not adjusted for planned GPIIb/IIIa inhibitor use or ACT). Participants who presented in the catheterization laboratory and who were receiving commercially available fondaparinux prescribed for the initial treatment of UA/NSTEMI may have been considered for randomization.
  Arms: Open label fondaparinux background and low dose UFH
Drug: Open label fondaparinux — Open-label fondaparinux syringes pre-filled with 2.5 mg, administered s.c. once daily for up to 8 days or hospital discharge, whichever was earlier, for those participants not indicated for PCI and not randomized
  Arms: Open label fondapaparinux

SUMMARY:
The purpose of this study is to compare the safety of two different dose regimens of unfractionated heparin (UFH) during a percutaneous coronary intervention (PCI) procedure in patients with UA (unstable angina)/NSTEMI (non ST segment elevation myocardial infarction) who have been initially treated with fondaparinux.

DETAILED DESCRIPTION:
Subjects presenting at hospital with suspected UA or NSTEMI and who are likely to undergo angiography (ideally within 72 hours) will be assessed for eligibility and consented. Suitable subjects will be enrolled and commence treatment with open-label fondaparinux, 2.5 milligram (mg), subcutaneous (s.c.), once daily. Following angiography subjects indicated for PCI and meeting the additional requirements for randomization will be randomised to receive one of two dose regimens of UFH either standard dose or low dose immediately prior to the PCI procedure. Post-PCI, therapy with fondaparinux (2.5 mg, s.c.) may be resumed at the investigator's discretion for up to a maximum of 8 days or hospital discharge, whichever is earlier.

Subjects not indicated for PCI, will continue treatment with fondaparinux, 2.5mg, s.c, once daily for up to 8 days or hospital discharge, whichever is earlier.

All subjects will be followed up for 30 days after randomization/angiography.

ELIGIBILITY:
The following are inclusion and exclusion criteria for enrollment in the study:

Inclusion Criteria:

* Presenting or admitted to hospital with symptoms suspected to represent UA or NSTEMI, i.e., clinical history consistent with new onset, or a worsening pattern of, characteristic ischemic chest pain or ischemic symptoms occurring at rest or with minimal activity (lasting longer than 5 minutes or requiring sublingual nitro-glycerine for relief of the pain).
* Available to be enrolled within 48 hours of the onset of the most recent episode of symptoms.
* Planned coronary angiography, with PCI if indicated, within 72 hours of enrollment where possible.
* At least two of the three following additional criteria:
* Age greater than or equal to 60 years
* Troponin T or I or CK-MB above the upper limit of normal for the local institution;
* Electrocardiogram (ECG) changes compatible with ischemia, i.e., ST depression at least 1 mm in 2 contiguous leads or T wave inversion > 3 mm or any dynamic ST shift or transient ST elevation.
* Written informed consent dated and signed

Exclusion Criteria:

* Age < 21 years.
* Any contraindication to UFH or fondaparinux
* Contraindication for angiography or PCI at baseline
* Subjects requiring urgent (<120 minutes) coronary angiography as characterized by those with:
* refractory or recurrent angina associated with dynamic ST-deviation
* heart failure
* life-threatening arrhythmias
* hemodynamic instability
* Subjects already receiving treatment with enoxaparin (or other LMWH), bivalirudin or UFH for treatment of the qualifying events unless the last administered (intravenous(i.v.) or s.c.) dose was:
* ≥ 8 hours for low molecular weight heparin (LMWH)
* ≥60 minutes for bivalirudin
* ≥90 minutes for unfractionated heparin (UFH)
* Hemorrhagic stroke within the last 12 months.
* Indication for anti-coagulation other than acute coronary syndrome (ACS) during the index hospitalization.
* Pregnancy or women of childbearing potential who are not using an effective method of contraception.
* Co-morbid condition with life expectancy less than 6 months.
* Currently receiving an experimental pharmacological agent.
* Revascularization procedure already performed for the qualifying event.
* Severe renal insufficiency (i.e., estimated creatinine clearance <20 ml/min)

Following angiography and confirmation that the subject is to undergo PCI, the subject must also meet all of the following additional criteria in order to be randomised:

* Subjects will have received at least 1 dose of open-label fondaparinux
* The most recent dose of open-label fondaparinux will not have been more than 24 hours before the start of the PCI procedure.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3235 (Actual)
Dates: Start 2009-02; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (164):
- United States (4):
  - GSK Investigational Site, Ocala, Florida
  - GSK Investigational Site, Albuquerque, New Mexico
  - GSK Investigational Site, Syracuse, New York
  - GSK Investigational Site, Dallas, Texas
- Argentina (11):
  - GSK Investigational Site, Adrogué, Buenos Aires
  - GSK Investigational Site, Bahía Blanca, Buenos Aires
  - GSK Investigational Site, La Plata, Buenos Aires
  - GSK Investigational Site, Merlo, Buenos Aires
  - GSK Investigational Site, Quilmes, Buenos Aires
  - GSK Investigational Site, Rosario, Buenos Aires
  - GSK Investigational Site, Corrientes, Corrientes Province
  - GSK Investigational Site, Rosario, Santa Fe Province
  - GSK Investigational Site, Santa Fe, Santa Fe Province
  - GSK Investigational Site, Buenos Aires
  - GSK Investigational Site, San Miguel de Tucumán
- Brazil (7):
  - GSK Investigational Site, Campina Grande do Sul, Paraná
  - GSK Investigational Site, Curitiba, Paraná
  - GSK Investigational Site, Porto Alegre, Rio Grande do Sul
  - GSK Investigational Site, Blumenau, Santa Catarina
  - GSK Investigational Site, Campinas, São Paulo
  - GSK Investigational Site, Marília, São Paulo
  - GSK Investigational Site, São José do Rio Preto, São Paulo
- Bulgaria (2):
  - GSK Investigational Site, Plovdiv
  - GSK Investigational Site, Sofia
- Canada (7):
  - GSK Investigational Site, Calgary, Alberta
  - GSK Investigational Site, Hamilton, Ontario
  - GSK Investigational Site, London, Ontario
  - GSK Investigational Site, Toronto, Ontario
  - GSK Investigational Site, Chicoutimi, Quebec
  - GSK Investigational Site, Montreal, Quebec
  - GSK Investigational Site, Québec, Quebec
- Czechia (7):
  - GSK Investigational Site, Brno
  - GSK Investigational Site, Hradec Králové
  - GSK Investigational Site, Karlovy Vary
  - GSK Investigational Site, Pilsen
  - GSK Investigational Site, Prague
  - GSK Investigational Site, Ústí nad Labem
  - GSK Investigational Site, Zlín
- France (10):
  - GSK Investigational Site, Besançon
  - GSK Investigational Site, Caen
  - GSK Investigational Site, Créteil
  - GSK Investigational Site, Dijon
  - GSK Investigational Site, Marseille
  - GSK Investigational Site, Montfermeil
  - GSK Investigational Site, Paris
  - GSK Investigational Site, Rouen
  - GSK Investigational Site, Toulouse
  - GSK Investigational Site, Tours
- Germany (32):
  - GSK Investigational Site, Heidelberg, Baden-Wurttemberg
  - GSK Investigational Site, Heidenheim, Baden-Wurttemberg
  - GSK Investigational Site, Bad Tölz, Bavaria
  - GSK Investigational Site, Dachau, Bavaria
  - GSK Investigational Site, Erlangen, Bavaria
  - GSK Investigational Site, Simbach A. Inn, Bavaria
  - GSK Investigational Site, Bernau bei Berlin, Brandenburg
  - GSK Investigational Site, Cottbus, Brandenburg
  - GSK Investigational Site, Bremen, City state Bremen
  - GSK Investigational Site, Hamburg, Hamburg
  - GSK Investigational Site, Kassel, Hesse
  - GSK Investigational Site, Langen, Hesse
  - GSK Investigational Site, Rüsselsheim am Main, Hesse
  - GSK Investigational Site, Bad Rothenfelde, Lower Saxony
  - GSK Investigational Site, Göttingen, Lower Saxony
  - GSK Investigational Site, Rostock, Mecklenburg-Vorpommern
  - GSK Investigational Site, Bonn, North Rhine-Westphalia
  - GSK Investigational Site, Cologne, North Rhine-Westphalia
  - GSK Investigational Site, Herford, North Rhine-Westphalia
  - GSK Investigational Site, Mönchengladbach, North Rhine-Westphalia
  - GSK Investigational Site, Neuss, North Rhine-Westphalia
  - GSK Investigational Site, Witten, North Rhine-Westphalia
  - GSK Investigational Site, Mainz, Rhineland-Palatinate
  - GSK Investigational Site, Homburg, Saarland
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Leipzig, Saxony
  - GSK Investigational Site, Halle, Saxony-Anhalt
  - GSK Investigational Site, Quedlinburg, Saxony-Anhalt
  - GSK Investigational Site, Lübeck, Schleswig-Holstein
  - GSK Investigational Site, Neumünster, Schleswig-Holstein
  - GSK Investigational Site, Berlin, State of Berlin
  - GSK Investigational Site, Erfurt, Thuringia
- Greece (3):
  - GSK Investigational Site, Athens
  - GSK Investigational Site, Ioannina
  - GSK Investigational Site, Rio- Patras
- Hungary (6):
  - GSK Investigational Site, Balatonfüred
  - GSK Investigational Site, Budapest
  - GSK Investigational Site, Debrecen
  - GSK Investigational Site, Miskolc
  - GSK Investigational Site, Pécs
  - GSK Investigational Site, Zalaegerszeg
- India (10):
  - GSK Investigational Site, Ahmedabad
  - GSK Investigational Site, Bandra, Mumbai
  - GSK Investigational Site, Bangalore
  - GSK Investigational Site, Dhantoli, Nagpur
  - GSK Investigational Site, Jaipur
  - GSK Investigational Site, Lucknow
  - GSK Investigational Site, New Delhi
  - GSK Investigational Site, Pune
  - GSK Investigational Site, Secunderabad
  - GSK Investigational Site, Vadodara
- Italy (12):
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Ferrara, Emilia-Romagna
  - GSK Investigational Site, Udine, Friuli Venezia Giulia
  - GSK Investigational Site, Cremona, Lombardy
  - GSK Investigational Site, Mantova, Lombardy
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pavia, Lombardy
  - GSK Investigational Site, Rozzano (Mi), Lombardy
  - GSK Investigational Site, Novara, Piedmont
  - GSK Investigational Site, Sassari, Sardinia
  - GSK Investigational Site, Lucca, Tuscany
  - GSK Investigational Site, Perugia, Umbria
- Netherlands (3):
  - GSK Investigational Site, Eindhoven
  - GSK Investigational Site, Nieuwegein
  - GSK Investigational Site, Rotterdam
- Poland (15):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Bytom
  - GSK Investigational Site, Częstochowa
  - GSK Investigational Site, Dąbrowa Górnicza
  - GSK Investigational Site, Gdansk
  - GSK Investigational Site, Gdynia
  - GSK Investigational Site, Koszalin
  - GSK Investigational Site, Krakow
  - GSK Investigational Site, Lubin
  - GSK Investigational Site, Radom
  - GSK Investigational Site, Torun
  - GSK Investigational Site, Warsaw
  - GSK Investigational Site, Wałbrzych
  - GSK Investigational Site, Wroclaw
  - GSK Investigational Site, Włocławek
- Russia (11):
  - GSK Investigational Site, Barnaul
  - GSK Investigational Site, Kemerovo
  - GSK Investigational Site, Krasnodar
  - GSK Investigational Site, Moscow
  - GSK Investigational Site, Novosibirsk
  - GSK Investigational Site, Perm
  - GSK Investigational Site, Saint Petersburg
  - GSK Investigational Site, St'Petersburg
  - GSK Investigational Site, Tomsk
  - GSK Investigational Site, Voronezh
  - GSK Investigational Site, Yaroslavl
- South Korea (8):
  - GSK Investigational Site, Busan
  - GSK Investigational Site, Daejeon
  - GSK Investigational Site, Gangnam-gu, Seoul
  - GSK Investigational Site, Goyang-si, Gyeonggi-do
  - GSK Investigational Site, Gwangju
  - GSK Investigational Site, Gyeonggi-do
  - GSK Investigational Site, Jeonju-si, Jeollabuk-Do
  - GSK Investigational Site, Seoul
- Spain (10):
  - GSK Investigational Site, Alicante
  - GSK Investigational Site, Galdakao
  - GSK Investigational Site, León
  - GSK Investigational Site, Madrid
  - GSK Investigational Site, Málaga
  - GSK Investigational Site, Oviedo
  - GSK Investigational Site, Palma de Mallorca
  - GSK Investigational Site, Santiago de Compostela
  - GSK Investigational Site, Seville
  - GSK Investigational Site, Vigo/Pontevedra
- United Kingdom (6):
  - GSK Investigational Site, Birmingham
  - GSK Investigational Site, Bristol
  - GSK Investigational Site, Dundee
  - GSK Investigational Site, Edinburgh
  - GSK Investigational Site, Southampton
  - GSK Investigational Site, Tooting, London

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] FUTURA/OASIS-8 Trial Group; Steg PG, Jolly SS, Mehta SR, Afzal R, Xavier D, Rupprecht HJ, Lopez-Sendon JL, Budaj A, Diaz R, Avezum A, Widimsky P, Rao SV, Chrolavicius S, Meeks B, Joyner C, Pogue J, Yusuf S. Low-dose vs standard-dose unfractionated heparin for percutaneous coronary intervention in acute coronary syndromes treated with fondaparinux: the FUTURA/OASIS-8 randomized trial. JAMA. 2010 Sep 22;304(12):1339-49. doi: 10.1001/jama.2010.1320. Epub 2010 Aug 31. PMID 20805623
- [Derived] Ducrocq G, Jolly S, Mehta SR, Rao SV, Patel T, Moreno R, Gao P, Steg PG. Activated clotting time and outcomes during percutaneous coronary intervention for non-ST-segment-elevation myocardial infarction: insights from the FUTURA/OASIS-8 Trial. Circ Cardiovasc Interv. 2015 Apr;8(4):e002044. doi: 10.1161/CIRCINTERVENTIONS.114.002044. PMID 25873729
- [Derived] Steg PG, Mehta S, Jolly S, Xavier D, Rupprecht HJ, Lopez-Sendon JL, Chrolavicius S, Rao SV, Granger CB, Pogue J, Laing S, Yusuf S. Fondaparinux with UnfracTionated heparin dUring Revascularization in Acute coronary syndromes (FUTURA/OASIS 8): a randomized trial of intravenous unfractionated heparin during percutaneous coronary intervention in patients with non-ST-segment elevation acute coronary syndromes initially treated with fondaparinux. Am Heart J. 2010 Dec;160(6):1029-34, 1034.e1. doi: 10.1016/j.ahj.2010.07.037. PMID 21146654
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Clinical Study Report: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: 108888 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: All participants (par.) received open-label (OL) fondaparinux (fond.). Par. indicated for percutaneous coronary intervention (PCI) were randomized to low- or standard-dose unfractionated heparin during PCI. Post-PCI, par. could resume OL fond. Par. not indicated for PCI weren't randomized and continued OL fond.
Groups:
- Open-label Fondaparinux 2.5 mg: Open-label (OL) fondaparinux syringes pre-filled with 2.5 milligrams (mg), administered subcutaneously (s.c.) once daily for up to 8 days or hospital discharge, whichever was earlier, for those participants not indicated for percutaneous coronary intervention (PCI) and not randomized
- OL Fondaparinux Background + Low Dose UFH During PCI: OL fondaparinux syringes pre-filled with 2.5 mg, administered s.c. once daily for up to 8 days or hospital discharge, whichever was earlier. Participants indicated for PCI were randomized to receive adjunctive blinded low-dose unfractionated heparin (UFH) (50 units/kilogram [U/kg], which was not adjusted for planned glycoprotein [GP] IIb/IIIa use or activated clotting time [ACT]). Participants who presented in the catheterization laboratory and who were receiving commercially available fondaparinux prescribed for the initial treatment of unstable angina/non-ST segment elevation myocardial infarction (UA/NSTEMI) may have been considered for randomization.
- OL Fondaparinux Background + Standard Dose UFH During PCI: OL fondaparinux syringes pre-filled with 2.5 mg, administered s.c. once daily for up to 8 days or hospital discharge, whichever was earlier. Participants indicated for PCI were randomized to receive adjunctive blinded standard dose UFH (based on planned GPIIb/IIIa inhibitor use: 60 U/kg; no planned use: 85 U/kg and adjusted based on ACT [maximum two additional bolus doses]). Participants who presented in the catheterization laboratory and who were receiving commercially available fondaparinux prescribed for the initial treatment of UA/NSTEMI may have been considered for randomization.
Period: Overall Study
Arm/Group | Open-label Fondaparinux 2.5 mg | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Started | 1209 | 1024 | 1002
Completed | 754 | 684 | 663
Not Completed | 455 | 340 | 339
Not completed — Adverse Event | 9 | 7 | 6
Not completed — Physician Decision | 304 | 271 | 255
Not completed — Withdrawal by Subject | 1 | 7 | 5
Not completed — Bleeding Event | 11 | 16 | 21
Not completed — Required Protocol-prohibited Therapy | 17 | 5 | 7
Not completed — Qualifying Condition Not Present | 29 | 14 | 16
Not completed — Verbatim Reason on the Case Report Form | 74 | 20 | 29
Not completed — Did Not Receive Study Drug | 10 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Open-label Fondaparinux 2.5 mg | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI | Total
Number analyzed (Participants) | 1209 | 1024 | 1002 | 3235
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.8 (11.07) | 65.3 (11.25) | 65.5 (11.10) | 65.5 (11.14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 486 | 335 | 316 | 1137
  Male | 723 | 689 | 686 | 2098
Race/Ethnicity, Customized [Number; unit: participants] — CRF, case report form.
  participants
    South Asian | 249 | 151 | 150 | 550
    Other Asian | 63 | 61 | 61 | 185
    Arab | 3 | 5 | 3 | 11
    Black African | 4 | 1 | 3 | 8
    European | 830 | 768 | 749 | 2347
    Native Latin | 57 | 37 | 33 | 127
    Other - verbatim reason collected on the CRF | 2 | 1 | 2 | 5
    Missing | 1 | 0 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Composite of Major Bleeding, Minor Bleeding, or Major Vascular Access Site Complications During the Peri-PCI Period
Description: The peri-percutaneous coronary intervention (peri-PCI) period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Major and minor bleeding events were adjudicated by a blinded central independent adjudication committee (CIAC). Major vascular access site complications comprised large hematoma, pseudoaneurysm requiring treatment, aterio-venous fistula, or other vascular procedures related to the access site.
Time Frame: Peri-PCI Period: occurred at randomization (from randomization to 48 hours after end of PCI procedure, typically 49 hours total)
Population: Intent-to-Treat (ITT) Population: all randomized participants
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants | 48 | 58
Statistical Analysis 1: Comparison: OL Fondaparinux Background + Low Dose UFH During PCI vs OL Fondaparinux Background + Standard Dose UFH During PCI; Test type: Superiority or Other; p = 0.267, Regression, Logistic; Odds Ratio (OR) = 0.80, 95% CI 2-sided [0.54 to 1.19]

2. Secondary Outcome: Number of Participants With Composite of Major Bleeding During the Peri-PCI Period, With Death, MI, or TVR at Day 30
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Assessment of death, myocardial infarction (MI) and target vessel revascularisation (TVR) was performed at Day 30. Major bleeding, MI and TVR were adjudicated by a blinded CIAC.
Time Frame: Peri-PCI period for major bleeding (during the time from randomization up to 48 hours after the end of PCI [typically 49 hours total] ) and from randomization up to Day 30 for death, MI, or TVR
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants | 59 | 39

3. Secondary Outcome: Number of Participants With Major Bleeding During the Peri-PCI Period
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Major bleeding, MI and TVR were adjudicated by a blinded CIAC.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants | 14 | 12

4. Secondary Outcome: Number of Participants With Minor Bleeding During the Peri-PCI Period
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Minor bleeding events were adjudicated by a blinded CIAC.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants | 7 | 17

5. Secondary Outcome: Number of Participants With Major Vascular Access Site Complications During the Peri-PCI Period
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Major vascular access site complications included: large hematoma, pseudoaneurysm requiring treatment, arterio-venous fistula, or other vascular procedures related to the access site.
Time Frame: as for outcome 1
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants | 33 | 43

6. Secondary Outcome: Number of Participants With Major PCI-related Procedural Complications
Description: Major PCI-related procedural complications included: abrupt vessel closure, a new angiographic filling defect representing either angiographic thrombus or major dissection with reduced flow, no-reflow phenomenon, or catheter-related thrombus. Investigator reports of catheter-related thrombus were defined as suspected catheter-related thrombus events, and were adjudicated by a blinded CIAC.
Time Frame: During PCI procedure: immediately after randomization (approximately 10-75 minutes)
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants
  Abrupt Vessel Closure | 10 | 17
  New Angiographic Thrombus | 11 | 8
  Suspected Catheter-related Thrombus | 4 | 3
  Catheter-related Thrombus-Adjudicated | 4 | 1
  No-reflow Phenomenon | 20 | 22
  New Major Dissection with Reduced Flow | 10 | 10

7. Secondary Outcome: Number of Participants With Composite of Death, MI or TVR During the Peri-PCI Period and at Day 30
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Assessment of composite of death, MI, or TVR was performed both during the peri-PCI period and at Day 30. MI and TVR events were adjudicated by a blinded CIAC.
Time Frame: Peri-PCI (during the time from randomization up to 48 hours after the end of PCI, typically 49 hours total) and from randomization up to Day 30
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants
  Composite of death, MI, and TVR Peri-PCI | 23 | 19
  Composite of death, MI, and TVR at Day 30 | 46 | 29

8. Secondary Outcome: Number of Participants Experiencing Death, MI, TVR, Definite/Probable Stent Thrombosis, or Stroke, Assessed Separately During the Peri-PCI Period and at Day 30
Description: The peri-PCI period was defined as the period during the time from randomization up to 48 hours after the end of the PCI procedure, typically 49 hours total. Assessment of death, MI, TVR, definite/probable stent thrombosis, or stroke was performed during the peri-PCI period and at Day 30. MI, TVR, definite/probable stent thrombosis, and stroke events were adjudicated by a blinded CIAC.
Time Frame: as for outcome 7
Population: ITT Population
Measure: Number; unit: participants
Arm/Group | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Number analyzed (Participants) | 1024 | 1002
participants
  Death during peri-PCI period | 1 | 2
  MI during peri-PCI period | 20 | 16
  TVR during peri-PCI period | 3 | 2
  Definite/Probable Stent Thrombosis during peri-PCI | 1 | 2
  Stroke during peri-PCI | 3 | 5
  Death at Day 30 | 8 | 6
  MI at Day 30 | 31 | 25
  TVR at Day 30 | 9 | 3
  Definite/Probable Stent Thrombosis at Day 30 | 12 | 5
  Stroke at Day 30 | 5 | 5

ADVERSE EVENTS:
Time Frame: Adverse events (AEs) and serious adverse events (SAEs) were collected from the start of fondaparinux until the follow-up at 30 days after randomization or angiography.
Description: Per the protocol, study outcome events (including bleeding, death, myocardial infarction [MI] and stroke, and other disease-related events) were not to be reported as AEs/SAEs.
Arm/Group | Open-label Fondaparinux 2.5 mg | OL Fondaparinux Background + Low Dose UFH During PCI | OL Fondaparinux Background + Standard Dose UFH During PCI
Serious Adverse Events (participants affected / at risk) | 48/1209 | 28/1024 | 20/1002
Other Adverse Events (participants affected / at risk) | 117/1209 | 100/1024 | 113/1002
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Fondaparinux 2.5 mg (N=1209) | OL Fondaparinux Background + Low Dose UFH During PCI (N=1024) | OL Fondaparinux Background + Standard Dose UFH During PCI (N=1002)
Pneumonia (Infections and infestations) | 4 | 2 | 2
Postoperative wound infection (Injury, poisoning and procedural complications) | 3 | 0 | 0
Renal failure acute (Renal and urinary disorders) | 3 | 3 | 0
Brain neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 2 | 0 | 0
Nephropathy toxic (Renal and urinary disorders) | 2 | 6 | 2
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 1
Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 0
Septic shock (Infections and infestations) | 2 | 0 | 0
Transient ischemic attack (Nervous system disorders) | 2 | 0 | 0
Acidosis (Metabolism and nutrition disorders) | 1 | 0 | 0
Anemia of chronic disease (Blood and lymphatic system disorders) | 1 | 0 | 0
Anal abscess (Infections and infestations) | 1 | 0 | 0
Aortic dissection (Vascular disorders) | 1 | 1 | 1
Atrial thrombosis (Cardiac disorders) | 1 | 0 | 0
Cholangitis (Hepatobiliary disorders) | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 1 | 0 | 0
Colitis ischaemic (Gastrointestinal disorders) | 1 | 0 | 0
Contrast media reaction (Injury, poisoning and procedural complications) | 1 | 0 | 1
Deep vein thrombosis (Vascular disorders) | 1 | 1 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0
Extremity necrosis (Vascular disorders) | 1 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 0
Gastroenteritis viral (Infections and infestations) | 1 | 0 | 0
Hepatic encephalophathy (Nervous system disorders) | 1 | 0 | 0
Hepatic enzyme increased (Investigations) | 1 | 0 | 0
Hepatic neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Impaired healing (General disorders) | 1 | 0 | 0
Intestinal ischemia (Gastrointestinal disorders) | 1 | 0 | 0
Lower respiratory tract infection (Infections and infestations) | 1 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Multiple myeloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Esophageal adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Esophagitis (Gastrointestinal disorders) | 1 | 0 | 0
Pericardial effusion (Cardiac disorders) | 1 | 0 | 0
Post procedural infection (Infections and infestations) | 1 | 0 | 0
Postoperative wound complication (Injury, poisoning and procedural complications) | 1 | 0 | 0
Renal artery stenosis (Renal and urinary disorders) | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0
Sepsis (Infections and infestations) | 1 | 0 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 1 | 2
Renal failure (Renal and urinary disorders) | 1 | 0 | 3
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 1
Arthritis bacterial (Infections and infestations) | 0 | 0 | 1
Bronchopneumonia (Infections and infestations) | 0 | 1 | 0
Cardiac tamponade (Cardiac disorders) | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0
Cholecystitis infective (Infections and infestations) | 0 | 0 | 1
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Colon cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Fecaloma (Gastrointestinal disorders) | 0 | 1 | 0
Hemolytic anemia (Blood and lymphatic system disorders) | 0 | 1 | 0
Hypertension (Vascular disorders) | 0 | 1 | 0
Neoplasm prostate (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0
Esophageal spasm (Gastrointestinal disorders) | 0 | 1 | 0
Pancreatic carcinoma metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1
Platelet count decreased (Investigations) | 0 | 0 | 1
Pleural hemorrhage (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1
Pyelonephritis acute (Infections and infestations) | 0 | 0 | 1
Urethral stenosis (Renal and urinary disorders) | 0 | 1 | 0
Urosepsis (Infections and infestations) | 0 | 1 | 0
Vascular access complication (Injury, poisoning and procedural complications) | 0 | 1 | 0
Vascular encephalopathy (Nervous system disorders) | 0 | 0 | 1
Vascular pseudoaneurysm (Injury, poisoning and procedural complications) | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 0.5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Open-label Fondaparinux 2.5 mg (N=1209) | OL Fondaparinux Background + Low Dose UFH During PCI (N=1024) | OL Fondaparinux Background + Standard Dose UFH During PCI (N=1002)
Headache (Nervous system disorders) | 18 | 24 | 28
Gastritis (Gastrointestinal disorders) | 15 | 0 | 2
Urinary tract infection (Infections and infestations) | 15 | 5 | 5
Asthenia (General disorders) | 13 | 7 | 3
Pyrexia (General disorders) | 13 | 11 | 16
Post procedural discharge (Injury, poisoning and procedural complications) | 11 | 9 | 15
Constipation (Gastrointestinal disorders) | 10 | 5 | 8
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 7 | 1
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 3
Carotid artery stenosis (Nervous system disorders) | 7 | 7 | 4
Hypercholesterolemia (Metabolism and nutrition disorders) | 7 | 3 | 5
Hypotension (Vascular disorders) | 7 | 6 | 10
Nausea (Gastrointestinal disorders) | 7 | 4 | 5
Vomiting (Gastrointestinal disorders) | 6 | 9 | 5
Dizziness (Nervous system disorders) | 5 | 11 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 9 | 7
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 10
Non-cardiac chest pain (General disorders) | 4 | 1 | 6
Hematoma (Vascular disorders) | 2 | 6 | 3
Nasopharyngitis (Infections and infestations) | 1 | 2 | 7
Hypertension (Vascular disorders) | 2 | 0 | 7
Insomnia (Psychiatric disorders) | 2 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.